CLINICAL TRIAL: NCT04186585
Title: Recommended Dose Estimation of BP-C2 in Patients With Prostate Cancer: A Phase I Dose-finding Study.
Brief Title: Recommended Dose Estimation of BP-C2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Meddoc (Other)
Collaborators: Meabco A/S (Industry)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor, Meddoc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PrCa-BPC2/I
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: BP-C2; Dose respons; Prostate Cancer; Hormon terapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Within-patient, 3-level Response Surface Pathway (RSP) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First design level (Experimental): All the 8 patients receives a daily oral dose of BP-C2 in ml equals the body weight divided by 5 for 4 weeks. This represents 15 ml for a patient of 75 kg
  Interventions: Drug: BP-C2
- Second design level (Experimental): Based on the results from the first design level, the daily BP-C2 dose will individually be increased by a factor of 1.4 or 1.2 in case of none or mild toxicity increase. If moderate or severe increase in toxicity is observed, the individual dose will be reduced by 0.8 or 0.6, respectively. Duration of the treatment is 4 weeks
  Interventions: Drug: BP-C2
- Third design level (Experimental): Based on the results from the second design level, the daily BP-C2 dose will individually be increased in case of none or mild toxicity increase and reduced if moderate or severe increase in toxicity is observed. Duration of the treatment is 4 weeks
  Interventions: Drug: BP-C2

INTERVENTIONS:
Drug: BP-C2 — Oral daily intake
  Other Names: Ammonium molybdate complexed with a lignin-derived polymer containing benzene polycarboxylic acids

SUMMARY:
The aim is to estimate an oral administered recommended dose of BP-C2 in addition to hormone treatment of prostate cancer.

The study population consists of prostatic cancer patients between 18 and 80 years of age undergoing hormonal treatment. Four patients will be recruited consecutively from each of two participating hospital.

The study will be performed as an open, one-dimensional multi-center trial with a 3-level within-patient Response Surface Pathway (RSP) design.

DETAILED DESCRIPTION:
Patients who seem to fulfil the inclusion without the exclusion criteria for the study will enter a screening phase of seven days. During this period, a clinical investigation will be performed, blood sample collected and prostate specific antigen (PSA) measured. The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity. Additionally, the quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be used. Both CTCAE and QoL will be recorded initially as individual baseline values. The trial treatment will start at the end of the screening period, denoted as Day 0, and the patients receiving study identification numbers.

BP-C2 will be administered orally once per day and the dose-window set to 0.33 - 1.67 mg/kg body weight (bw). For an average patient of 75 kg this represents 5 - 25 ml. The starting dose will be 1.0 mg/kg bw representing 15 ml for an average patient. All the eight participating patients will receive the daily starting dose of 1.0 mg/kg bw for four weeks at the first design-level. The study consists of three design-levels, each of four weeks duration. CTCAE and QoL registration will be performed after two and four weeks at each design-level. In case of life threatening, serious adverse events, or occurrence of unacceptable side effects related to the trial substance, the treatment will be stopped.

The CTCAE results are shown in the two variables "Sum CTCAE score" and "Max CTCAE". The tolerability classification used in the study design is based on the Max score as: "0=none", "1=mild", "2= moderate", "3= severe", "4= Life threatening" and "5= death". The change in the Max score from the study baseline to four weeks of BP-C2 treatment [4 weeks - baseline] are classified as "0= unchanged or reduced", "1=small increase", "2= moderate increase", "3= severe increase" and "4= life-threatening increase". In case the change in the Max score is classified as 0 or 1, the dose to be used for the patient at the next design level will be increased. If the change is 2 or 3, the dose will be reduced. Termination of the study occurs if the change in the Max score is 4 or larger. The size of the dose escalation or de-escalation will be calculated in accordance with the Response Surface Pathway (RSP) procedure depending on the change in Max CTCAE score from baseline to the end of each design-level. Based on the results obtained after four weeks of treatment at one design level, the dose to be used at the next design level will be individually calculated.

Each patient will be followed up four weeks after end of treatment with final CTCAE and QoL registration.

The CTCAE related variables are the main variables in this study. The secondary variables are the QoL variables EQ index and EQ-VAS.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients between 18 and 80 years of age under hormonal treatment

Exclusion Criteria:

* Patients with expected survival time below 3 months
* Abnormal liver function classified as total bilirubin >34 µmol/l or ALAT > 3 times the upper normal range (ULN). In case of metastases in the liver, the ALAT limit for exclusion is set to 5 x ULN.
* Abnormal kidney function defined by serum creatinine >120 µmol/l.
* Patients with verified metastasis to the brain.
* Synchronous cancer except for non-melanoma skin cancer and early stage of cervical cancer.
* Clinically significant abnormal ECG.
* Under radiological therapy
* Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* Not able to understand information.
* Do not want or not able to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men due to the diagnos
Enrollment: 8 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Max CTCAE | Week 0
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Max CTCAE | Week 2
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Max CTCAE | Week 4
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Max CTCAE | Week 6
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Max CTCAE | Week 8
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Sum CTCAE score | Week 0
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Sum CTCAE score | Week 2
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Sum CTCAE score | Week 4
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Sum CTCAE score | Week 6
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Sum CTCAE score | Week 8
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Quality of Life questionnaire (EQ-5D-5L) | Week 0
  Five score levels: "Mobility", "Self-care","Usual activity", "Pain/Discomfort", "Anxiety/Depression" and "Overall daily health situation"
Quality of Life questionnaire (EQ-5D-5L) | Week 4
  Five score levels: "Mobility", "Self-care","Usual activity", "Pain/Discomfort", "Anxiety/Depression" and "Overall daily health situation"
Quality of Life questionnaire (EQ-5D-5L) | Week 8
  Five score levels: "Mobility", "Self-care","Usual activity", "Pain/Discomfort", "Anxiety/Depression" and "Overall daily health situation"
PSA | Week 0
  Prostate marker
PSA | Week 4
  Prostate marker
PSA | Week 8
  Prostate marker

CONTACTS AND LOCATIONS:
Overall Officials: Svein Aa Ingelholm, PhD, Study Chair — Meabco A/S
Locations (1):
- Meddoc, Skjetten, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
The data will be available for the study inverstigators, statistician and the data manager